CLINICAL TRIAL: NCT05035004
Title: The Effects of Post Aerobic Exercise Hot Water Immersion on Physiological and Perceptual Responses in Physically Inactive Middle-aged Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coventry University (Other)
Responsible Party: Principal Investigator, Charles Steward, Post Graduate Research Student in the Centre for Sport, Exercise and Life Sciences, Coventry University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: P97102
Record Dates: First submitted 2021-08-06; First posted 2021-09-05 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Healthy Aging
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Post exercise hot water immersion (Experimental): Moderate intensity cycling for 30 minutes, followed by a 10-minute transfer period and then 30 minutes of whole-body hot water immersion.
  Interventions: Device: Post exercise hot water immersion
- Exercise (Active Comparator): Moderate intensity cycling for 30 minutes.
  Interventions: Device: Exercise
- Hot water immersion (Active Comparator): Whole-body hot water immersion for 30 minutes, followed by a 10-minute transfer period and then an additional 30 minutes of whole-body hot water immersion.
  Interventions: Device: Hot water immersion

INTERVENTIONS:
Device: Post exercise hot water immersion — Participants will complete 30 minutes of cycling on a lode bicycle ergometer (50% of VO2max), followed by a 10-minute transfer period and then 30 minutes of whole-body hot water immersion in a hot tub (water temperature 40°C).
  Arms: Post exercise hot water immersion
Device: Exercise — Participants will complete 30 minutes of cycling on a lode bicycle ergometer (50% of VO2max).
  Arms: Exercise
Device: Hot water immersion — Participants will complete 30 minutes of whole-body hot water immersion in a hot tub (water temperature 40°C), followed by a 10-minute transfer period and then an additional 30 minutes of whole-body hot water immersion in a hot tub (water temperature 40°C).
  Arms: Hot water immersion

SUMMARY:
This study will investigate the effects of post moderate intensity aerobic exercise hot water immersion on physiological and perceptual responses in physically inactive middle-aged adults when compared to moderate intensity aerobic exercise and hot water immersion alone.

DETAILED DESCRIPTION:
A large number of middle aged adults do not achieve the minimum recommended amount of physical activity. This consequently increases the risk of cardiovascular disease and all-cause mortality. Although below the recommended physical activity guidelines, it is important to highlight that a considerable proportion of these individuals do take part in some form of physical activity within their weekly routines. Hence, identifying complementary therapies that can enhance the health benefits from smaller amounts of exercise are of great value for many physically inactive middle-aged adults.

An in increase in body temperature from a single session of passive heating has been shown to mimic many of the beneficial physiological responses of exercise, such as, an increase in heart rate, skin blood flow and an increase in circulating angiogenic factors. However, lab based studies often push participants to the limit of thermal tolerance which may reduce long term adherence in the real world. Therefore, this study will investigate whether the use of post exercise hot water immersion can prolong and / or intensify exercise mediated physiological responses that underpin health benefits, whilst also assessing the perceptual responses, in comparison to exercise and hot water immersion alone.

Through the use of a repeated measures design, participants will randomly take part in three conditions; 1) post exercise hot water immersion (30 minutes of moderate intensity cycling followed by 10 minutes of supine rest and 30 minutes of whole body hot water immersion at 40°C); 2) aerobic exercise (30 minutes of moderate intensity cycling followed by 10 minutes of supine rest and 30 minutes of seated rest at room temperature); 3) hot water immersion condition (30 minutes of whole body hot water immersion at 40°C followed by 10 minutes of supine rest and 30 minutes of whole body hot water immersion at 40°C). Each condition will be separated by a minimum of 1-week. Outcome measures will either be assessed at regular intervals or at 0, 30, 70 and 100 minute time points for each condition.

ELIGIBILITY:
Inclusion Criteria:

* Males and post menopausal females
* Aged between 40 - 60 years
* BMI of 18.5 - 34.9 kg/m2
* Over the last 6 months has participated in less than 150 mins of moderate intensity physical activity or 75 mins of vigorous activity or a combination of both, but takes part in some form of physical activity within their weekly routine.
* Maximal oxygen uptake categorised as 'fair' for a given age group.

Exclusion Criteria:

* Previous myocardial infarction or cerebrovascular event
* Any signs or symptoms of cardiovascular issues
* High blood pressure: SBP >180 mmHg and / or DBP >100 mmHg
* Orthostatic hypotension: Drop of SBP > 20mmHg and / or DBP >10 mmHg upon standing.
* Changed blood pressure medication in the 6-month period prior to the study
* Plan to change any form of relevant medication during study period
* Suffers from diabetes
* Suffers from severe asthma
* Currently have any infections or symptoms of an infection (e.g. COVID-19 etc)
* Suffers from a neurodegenerative disease
* Cannot understand and/or fully cooperate with the study protocol
* Exercise-limiting comorbidity (e.g. angina, chronic lung disease, arthritis etc)
* Severe peripheral neuropathy (cannot sense temperature)
* Current smoker or have stopped in the last 3 months
* Any skin conditions including ulcerations
* Exposed to high temperatures in the last 4-weeks (e.g. holiday, spa, sun beds etc)
* Use of antioxidant supplements in the last 6-weeks

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
Change in circulating plasma nitrite (pg/ml) | Measured at 0, 30, 70 and 100 minutes
  Venous blood sample
Change in brachial artery total shear rate (S-1) | Measured at 0, 30, 70 and 100 minutes
  Terason ultrasound recording of the brachial and superficial femoral artery
Change in brachial artery antegrade shear rate (S-1) | Measured at 0, 30, 70 and 100 minutes
  Terason ultrasound recording of the brachial and superficial femoral artery.
Change in brachial artery retrograde shear rate (S-1) | Measured at 0, 30, 70 and 100 minutes
  Terason ultrasound recording of the brachial and superficial femoral artery
Change in brachial artery diameter (mm) | Measured at 0, 30, 70 and 100 minutes
  Terason ultrasound recording of the brachial and superficial femoral artery
Change in brachial artery blood flow (ml/min) | Measured at 0, 30, 70 and 100 minutes
  Terason ultrasound recording of the brachial and superficial femoral artery.
Change in brachial artery compliance (μm/mmHg) | Measured at 0, 30, 70 and 100 minutes
  Terason ultrasound recording of the brachial artery. Brachial artery compliance will be calculated by using the change in blood volume and blood pressure
Change in systolic blood pressure (mmHg) | Measurements taken at 10 minute intervals up to 100 minutes
  Measured using an automated blood pressure cuff
Change in diastolic blood pressure (mmHg) | Measurements taken at 10 minute intervals up to 100 minutes
  Measured using an automated blood pressure cuff
Change in mean arterial pressure (mmHg) | Measurements taken at 10 minute intervals up to 100 minutes
  Measured using an automated blood pressure cuff. Mean arterial pressure will be calculated by using systolic and diastolic blood pressure
Change in pulse pressure (mmHg) | Measurements taken at 10 minute intervals up to 100 minutes
  Measured using an automated blood pressure cuff. Pulse pressure will be calculated using systolic and diastolic blood pressure

SECONDARY OUTCOMES:
Change in circulating serum Interleukin-6 (pg/ml) | Measured at 0, 30, 70 and 100 minutes
  Venous blood sample
Change in circulating serum Interleukin-10 (pg/ml) | Measured at 0, 30, 70 and 100 minutes
  Venous blood sample
Change in circulating serum Interleukin-8 (pg/ml) | Measured at 0, 30, 70 and 100 minutes
  Venous blood sample
Change in circulating serum Interleukin-1Ra (pg/ml) | Measured at 0, 30, 70 and 100 minutes
  Venous blood sample
Change in circulating serum Vascular endothelial growth factor (pg/ml) | Measured at 0, 30, 70 and 100 minutes
  Venous blood sample
Change in circulating serum Endothelin-1 (pg/ml) | Measured at 0, 30, 70 and 100 minutes
  Venous blood sample
Circulating serum Monocyte chemoattractant protein-1 (pg/ml) | Measured at 0, 30, 70 and 100 minutes
  Venous blood sample
Change in circulating serum Matrix metallopeptidase-2 (pg/ml) | Measured at 0, 30, 70 and 100 minutes
  Venous blood sample
Change in circulating serum Matrix metallopeptidase-9 (pg/ml) | Measured at 0, 30, 70 and 100 minutes
  Venous blood sample
Energy expenditure (kcal/h-1) | Gas measurements taken continually up to 70 minutes. Energy expenditure calculated from the 30 minutes of exercise, hot water immersion and/or rest periods.
  Measured initially by breath by breath analysis through the use of a Ultima and calculated via indirect calorimetry
Change in thermal comfort | Measured at 10 minute intervals up to 100 minutes
  Thermal comfort Likert scale from a positive score of +5 very comfortable (maximum) to a negative score of -5 very uncomfortable (minimum)
Change in thermal sensation | Measured at 10 minute intervals up to 100 minutes
  Thermal sensation Likert scale from +5 (maximum) hot to -5 cold (minimum)
Change in basic affect | Measured at 10 minute intervals up to 100 minutes
  Basic affect Likert scale from a positive score of +5 very good (maximum) to a negative score of -5 very bad (minimum)
Change in physical activity enjoyment scale | Measured ~12 minutes post intervention
  Feelings about exercise and / or passive heating on a Likert scale from a positive score of 1 (maximum) to a negative score of 7 (minimum)

OTHER OUTCOMES:
Change in rectal core temperature (°C) | Measurements taken at 10 minute intervals up to 100 minutes
  Measured using a rectal probe attached to a squirrel data logger
Change in forehead skin temperature (°C) | Measurements taken at 10 minute intervals up to 100 minutes
  Measured using skin thermistors attached to a squirrel data logger
Change in heart rate (bpm) | Measurements taken at 10 minute intervals up to 100 minutes
  Measured using a heart rate monitor
Change in plasma volume (%) | Measurements taken pre and immediately post intervention
  Measured by a capillary blood sample then calculating plasma volume via the hemoglobin and hematocrit

CONTACTS AND LOCATIONS:
Locations (1):
- Coventry University, Coventry, West Midlands, United Kingdom